CLINICAL TRIAL: NCT00630474
Title: Does Nasal Decongestion Improve Obstructive Sleep Apnea ?
Brief Title: Nasal Decongestion and Obstructive Sleep Apnea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Konrad E. Bloch, Professor, MD, University Hospital Zurich, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EK-825
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Obstructive Sleep Apnea Syndrome; Rhinitis
Keywords: sleep apnea, rhinitis
MeSH Terms: conditions — Sleep Apnea, Obstructive; Rhinitis; Sleep Apnea Syndromes | interventions — xylometazoline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): nasal application of xylometazoline
  Interventions: Drug: xylometazoline
- 2 (Placebo Comparator): nasal application of placebo
  Interventions: Drug: xylometazoline

INTERVENTIONS:
Drug: xylometazoline — xylometazoline (0.1 % solution, 3 drops, 0.15 mg) in each nostril
  Other Names: Otrivin

SUMMARY:
Whether impaired nasal breathing contributes to sleep related breathing disturbances has not been known. Therefore, the purpose of the study is to compare the effect of xylometazoline, a drug that decongests the nasal mucosa when applied locally, with placebo in terms of sleep and nocturnal breathing and daytime performance.

ELIGIBILITY:
Inclusion Criteria:

* Obstructive sleep apnea syndrome (excessive sleepiness, apnea/hypopnea index >10/h)
* Chronic nasal congestion (complaint of impaired nasal breathing that interfered with subjective sleep quality on at least 3 nights per week during at least the last 3 months)

Exclusion Criteria:

* Nasal surgery within the last 6 months
* Current treatment with nasal decongestants or topical steroids
* Sleep disorders other than obstructive sleep apnea
* Internal medical or psychiatric disorders that interfered with sleep

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-01; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
sleep related breathing disturbances sleep efficiency daytime sleepiness | at end of one week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Konrad E Bloch, MD, Study Chair — University Hospital, Zürich
Locations (2):
- Switzerland (2):
  - Pulmonary Division, University Hospital Zurich, Switzerland, Zurich
  - Pulmonary Division, University Hospital Zurich, Zurich

REFERENCES:
- [Result] Clarenbach CF, Kohler M, Senn O, Thurnheer R, Bloch KE. Does nasal decongestion improve obstructive sleep apnea? J Sleep Res. 2008 Dec;17(4):444-9. doi: 10.1111/j.1365-2869.2008.00667.x. Epub 2008 Aug 15. PMID 18710420